CLINICAL TRIAL: NCT01472510
Title: Ranibizumab in Residual Diabetic Macular Edema Following Previous Anti-VEGF Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vitreo-Retinal Associates, PC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27906
Record Dates: First submitted 2011-11-03; First posted 2011-11-16 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic; Macular; Edema; Ranibizumab; anti-VEGF
MeSH Terms: conditions — Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1:The PRN Group (Active Comparator): You will receive 6 monthly intravitreal injections of 0.5% Ranibizumab administered about every 28 days. It is possible you may receive additional injections into the study eye for the next six months if certain criteria is met.
  Interventions: Drug: Ranibizumab
- arm 2:The Monthly Group: (Active Comparator): You will receive 12 monthly intravitreal injections of 0.5% Ranibizumab administered every 28 days.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — A 0.5mg intravitreal injection of Ranibizumab will be administered to subjects. Subjects will receive 6 monthly consecutive ranibizumab injections. Study visits will be scheduled to occur every 28 days relative to the date of the first injection
  Other Names: lucentis
  Arms: Arm 1:The PRN Group
Drug: Ranibizumab — A 0.5mg intravitreal injection of Ranibizumab will be administered to subjects. Subjects will receive 12 monthly consecutive ranibizumab injections. Study visits will be scheduled to occur every 28 days relative to the date of the first injection
  Other Names: lucentis
  Arms: arm 2:The Monthly Group:

SUMMARY:
This study is designed to confirm that the investigational drug Ranibizumab given by injection into the eye is safe and effective to use in people with diabetic macular edema (DME).

DETAILED DESCRIPTION:
Ranibizumab works by blocking Vascular Endothelial Growth Factor (VEGF), a substance which is found in eyes with diabetic eye disease and which causes leakage from blood vessels. Several studies have suggested that eyes with DME may have very high levels of VEGF; therefore, Ranibizumab may be helpful in blocking VEGF and decreasing DME.

Ranibizumab has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of wet age-related macular degeneration (AMD) and Retinal Vein Occlusion at the dose amount of 0.5 mg. Ranibizumab has not been approved for use in subjects with DME.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:

  1. Age > 18 years
  2. Diagnosis of diabetes mellitus (type 1 or 2)
  3. Residual edema as determined by mean foveal thickness on Cirrus OCT > 300 microns and leakage seen on FA at baseline
  4. Clinical evidence of retinal thickening due to macular edema involving the center of the macula, associated with diabetic retinopathy.
  5. Previous history of at least 4 or more consecutive anti-VEGF intravitreal injections of Pegaptanib sodium or Bevacizumab (consecutive injections administered no more than 6 weeks apart in the last year) for the treatment of diabetic macular edema.
  6. Previous history of focal laser and/or intravitreal steroid injection for the treatment of diabetic macular edema.
  7. BCVA of 20/32-20/400 (ETDRS)
  8. Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

1. Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception. . The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
2. Participation in another ocular investigation or trial simultaneously.
3. Systemic use of anti-VEGF within 3 months prior to day 0.
4. Previous intravitreal ranibizumab within 3 months prior to day 0
5. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110)
6. Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism, drug abuse).
7. Evidence of vitreoretinal interface abnormality after ocular exam or OCT that may be contributing to the macular edema.
8. An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of subretinal fibrosis, ischemic maculopathy or geographic atrophy).
9. Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (e.g. AMD, uveitis, Irvine-Gass).
10. Evidence of active neovascularization of the iris or retina.
11. Evidence of central atrophy or fibrosis in the study eye.
12. Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
13. History of vitreous surgery in the study eye.
14. History of cataract surgery within 6 months of enrollment.
15. History of YAG capsulotomy within 2 months of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Acuity Scores at Month 12 Compared to Baseline | 12 months

SECONDARY OUTCOMES:
Resolution of residual edema compared to baseline as determined by mean foveal thickness on Cirrus OCT 300 microns at Month 6 and Month 12. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank J McCabe, M.D., Principal Investigator — Vitreo-Retinal Associates, PC; Marie V Lampson, Study Director — Vitreo-Retinal Associates, PC
Locations (1):
- Vitreo-Retinal Associates, PC, Worcester, Massachusetts, United States